CLINICAL TRIAL: NCT03629262
Title: Impact of Dexmedetomidine Supplemented Intravenous Analgesia on Postoperative Delirium and Long-term Outcomes in Elderly After Orthopedic Surgery: A Multicenter, Double-blinded, Randomized Controlled Trial
Brief Title: Dexmedetomidine Supplemented Intravenous Analgesia in Elderly After Orthopedic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-131; ChiCTR1800017182 (Registry Identifier: Chinese Clinical Trial Registry (www.chictr.org.cn))
Record Dates: First submitted 2018-08-08; First posted 2018-08-14 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Elderly; Orthopedic Surgery; Analgesia; Dexmedetomidine; Postoperative Delirium; Long-term Outcome
Keywords: Elderly; Orthopedic Surgery; Analgesia; Dexmedetomidine; Postoperative Delirium; Long-term Outcome
MeSH Terms: conditions — Agnosia; Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Experimental): For patients in the dexmedetomidine group, postoperative analgesia is provided in the form of patient-controlled intravenous analgesia. The formula contains a mixture of sufentanil (1.25 ug/ml) and dexmedetomidine (1.25 ug/ml), diluted with normal saline to a total volume of 160 ml. The analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with a patient-controlled bolus of 2 ml each time and a lockout interval of 8 minutes.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): For patients in the control group, postoperative analgesia is provided in the form of patient-controlled intravenous analgesia. The formula contains a mixture of placebo and sufentanil (1.25 ug/ml), diluted with normal saline to a total volume of 160 ml. The analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with a patient-controlled bolus of 2 ml each time and a lockout interval of 8 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Patients in this group receive patient-controlled intravenous analgesia for 1-3 days after surgery. The formula is a mixture of dexmedetomidine (1.25 ug/ml) and sufentanil (1.25 ug/ml), diluted with normal saline to 160 ml. 5-HT3 receptor antagonist is added when necessary. The analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with a bolus dose of 2 ml at each time and a lockout interval of 8 minutes.
  Other Names: Sufentanil analgesia
  Arms: Dexmedetomidine group
Drug: Placebo — Patients in this group receive patient-controlled intravenous analgesia for 1-3 days after surgery. The formula is a mixture of placebo and sufentanil (1.25 ug/m), diluted with normal saline to 160 ml. 5-HT3 receptor antagonist is added when necessary. The analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with a bolus dose of 2 ml at each time and a lockout interval of 8 minutes.
  Other Names: Sufentanil analgesia
  Arms: Control group

SUMMARY:
Delirium is common in the elderly after orthopedic surgery and is associated with worse outcomes. The investigators hypothesize that, for elderly patients after orthopedic surgery, dexmedetomidine supplemented intravenous analgesia can reduce the incidence of delirium and improve the long-term outcomes.

DETAILED DESCRIPTION:
A growing number of elderly patients undergo orthopedic surgery each year. Delirium is a common complication in these patients after surgery and is associated with worse outcomes, including prolonged hospital stay, poor functional recovery, decreased cognitive function, increased health care costs, and elevated mortality rate. Previous studies showed that, for elderly patients admitted to the intensive care unit after non-cardiac surgery, low-dose dexmedetomidine infusion improved subjective sleep quality and reduced delirium early after surgery; it also increased survival up to 2 years and improved life quality in 3-year survivors. The investigators hypothesize that dexmedetomidine supplemented intravenous analgesia (in the form of patient-controlled analgesia) can also reduce delirium and improve long-term outcomes in elderly patients after orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years but < 90 years;
* Scheduled to undergo total knee/hip replacement surgery, or spinal surgery;
* Planned to use patient-controlled intravenous analgesia (PCIA) after surgery.

Exclusion Criteria:

* Refuse to participate in this study;
* Preoperative history of schizophrenia, epilepsy, Parkinsonism, or myasthenia gravis;
* Inability to communicate in the preoperative period because of coma, profound dementia or language barrier;
* Preoperative obstructive sleep apnea (diagnosed sleep apnea syndrome or a STOP-Bang score ≥3 combined with a serum bicarbonate ≥28 mmol/L);
* Sick sinus syndrome, severe sinus bradycardia (< 50 beats per minute), or second-degree or above atrioventricular block without pacemaker;
* Severe hepatic dysfunction (Child-Pugh class C);
* Severe renal dysfunction (requirement of renal replacement therapy before surgery);
* American Society of Anesthesiologists physical status >IV, or estimated survival ≤24 h.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 712 (Actual)
Dates: Start 2018-10-28 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium within the first 5 days after surgery | The first 5 days after surgery
  Incidence of delirium within the first 5 days after surgery

SECONDARY OUTCOMES:
Daily prevalence of delirium during the first 5 days after surgery | The first 5 days after surgery
  Daily prevalence of delirium during the first 5 days after surgery
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of non-delirium complications with 30 days after surgery | Up to 30 days after surgery
  Incidence of non-delirium complications with 30 days after surgery
All-cause 30-day mortality | Up to 30 days after surgery
  All-cause 30-day mortality
Quality of life of 30-day survivors | At 30 days after surgery
  Quality of life of 30-day survivors is assessed with World Health Organization Quality of Life brief version (WHOQOL-BREF), a 24-item questionnaire that provides assessments of the quality of life in physical, psychological, social relationship, and environmental domains. For each domain, the score ranges from 0 to 100, with higher score indicating better function.
Cognitive function of 30-day survivors | At 30 days after surgery
  Cognitive function of 30-day survivors is assessed with the modified Telephone Interview for Cognitive Status (TICS-m), a 12-item questionnaire that provides an assessment of global cognitive function by verbal communication via telephone. The score ranges from 0 to 48, with higher score indicating better function.
Agitation or sedation level during postoperative days 1-5 | The first 1-5 days after surgery
  Agitation or sedation level is assessed twice daily with the Richmond Agitation-Sedation Scale (RASS), of which the range is as follows: +4 (combative), +3 (very agitated), +2 (agitated), +1 (restless), 0 (alert and clam), -1 (drowsy), -2 (light sedation), -3 (moderate sedation), -4 (deep sedation), and -5 (unarousable).
Cumulative sufentanil consumption within 5 postoperative days | Up to 5 days after surgery
  Cumulative sufentanil consumption within 5 postoperative days
Pain severity during postoperative days 1-5 | The first 1-5 days after surgery
  Pain severity is assessed with twice daily the Numeric Rating Scale (NRS), an 11 point scale where 0=no pain and 10=the worst possible pain.
Subjective sleep quality during postoperative days 1-5 | The first 1-5 days after surgery
  Subjective sleep quality is assessed once daily with the Numeric Rating Scale (NRS), an 11 point scale where 0=the best sleep and 10=the worst sleep.
Overall survival for up to 3 years after surgery | Up to 3 years after surgery
  Time from surgery to all-cause death for up to 3 years after surgery.
Event-free survival for up to 3 years after surgery | Up to 3 years after surgery
  Time from surgery to new-onset diseases or all-cause death, whichever comes first. New-onset disease indicates those that required hospital admission and/or interventional procedure.
Quality of life in 1-，2- and 3-year survivors after surgery | At the end of the 1st, 2nd, and 3rd year after surgery
  Quality of life in 1-，2- and 3-year survivors is assessed with the WHOQOL-BREF, a 24-item questionnaire that provides assessments of the quality of life in physical, psychological, social relationship, and environmental domains. For each domain, the score ranges from 0 to 100, with higher score indicating better function.
Cognitive function in 1-，2- and 3-year survivors after surgery | At the end of the 1st, 2nd, and 3rd year after surgery
  Cognitive function in 1-，2- and 3-year survivors is assessed with the TICS-m, a 12-item questionnaire that provides an assessment of global cognitive function by verbal communication via telephone. The score ranges from 0 to 48, with higher score indicating better function.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dyer CB, Ashton CM, Teasdale TA. Postoperative delirium. A review of 80 primary data-collection studies. Arch Intern Med. 1995 Mar 13;155(5):461-5. doi: 10.1001/archinte.155.5.461. PMID 7864702
- [Background] McDaniel M, Brudney C. Postoperative delirium: etiology and management. Curr Opin Crit Care. 2012 Aug;18(4):372-6. doi: 10.1097/MCC.0b013e3283557211. PMID 22732435
- [Background] Mu DL, Wang DX, Li LH, Shan GJ, Li J, Yu QJ, Shi CX. High serum cortisol level is associated with increased risk of delirium after coronary artery bypass graft surgery: a prospective cohort study. Crit Care. 2010;14(6):R238. doi: 10.1186/cc9393. Epub 2010 Dec 30. PMID 21192800
- [Background] Shi CM, Wang DX, Chen KS, Gu XE. Incidence and risk factors of delirium in critically ill patients after non-cardiac surgery. Chin Med J (Engl). 2010 Apr 20;123(8):993-9. PMID 20497703
- [Background] Lat I, McMillian W, Taylor S, Janzen JM, Papadopoulos S, Korth L, Ehtisham A, Nold J, Agarwal S, Azocar R, Burke P. The impact of delirium on clinical outcomes in mechanically ventilated surgical and trauma patients. Crit Care Med. 2009 Jun;37(6):1898-905. doi: 10.1097/CCM.0b013e31819ffe38. PMID 19384221
- [Background] Quinlan N, Rudolph JL. Postoperative delirium and functional decline after noncardiac surgery. J Am Geriatr Soc. 2011 Nov;59 Suppl 2:S301-4. doi: 10.1111/j.1532-5415.2011.03679.x. PMID 22091577
- [Background] Lescot T, Karvellas CJ, Chaudhury P, Tchervenkov J, Paraskevas S, Barkun J, Metrakos P, Goldberg P, Magder S. Postoperative delirium in the intensive care unit predicts worse outcomes in liver transplant recipients. Can J Gastroenterol. 2013 Apr;27(4):207-12. doi: 10.1155/2013/289185. PMID 23616958
- [Background] Abelha FJ, Luis C, Veiga D, Parente D, Fernandes V, Santos P, Botelho M, Santos A, Santos C. Outcome and quality of life in patients with postoperative delirium during an ICU stay following major surgery. Crit Care. 2013 Oct 29;17(5):R257. doi: 10.1186/cc13084. PMID 24168808
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Van Rompaey B, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Elseviers M, Bossaert L. Long term outcome after delirium in the intensive care unit. J Clin Nurs. 2009 Dec;18(23):3349-57. doi: 10.1111/j.1365-2702.2009.02933.x. Epub 2009 Sep 4. PMID 19735334
- [Background] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966
- [Background] Stuck A, Clark MJ, Connelly CD. Preventing intensive care unit delirium: a patient-centered approach to reducing sleep disruption. Dimens Crit Care Nurs. 2011 Nov-Dec;30(6):315-20. doi: 10.1097/DCC.0b013e31822fa97c. PMID 21983504
- [Background] Siddiqi N, Harrison JK, Clegg A, Teale EA, Young J, Taylor J, Simpkins SA. Interventions for preventing delirium in hospitalised non-ICU patients. Cochrane Database Syst Rev. 2016 Mar 11;3(3):CD005563. doi: 10.1002/14651858.CD005563.pub3. PMID 26967259
- [Background] Kosar CM, Tabloski PA, Travison TG, Jones RN, Schmitt EM, Puelle MR, Inloes JB, Saczynski JS, Marcantonio ER, Meagher D, Reid MC, Inouye SK. EFFECT OF PREOPERATIVE PAIN AND DEPRESSIVE SYMPTOMS ON THE DEVELOPMENT OF POSTOPERATIVE DELIRIUM. Lancet Psychiatry. 2014 Nov;1(6):431-436. doi: 10.1016/S2215-0366(14)00006-6. PMID 25642413
- [Background] Halaszynski TM. Pain management in the elderly and cognitively impaired patient: the role of regional anesthesia and analgesia. Curr Opin Anaesthesiol. 2009 Oct;22(5):594-9. doi: 10.1097/ACO.0b013e32833020dc. PMID 19623056
- [Background] Brummel NE, Girard TD. Preventing delirium in the intensive care unit. Crit Care Clin. 2013 Jan;29(1):51-65. doi: 10.1016/j.ccc.2012.10.007. PMID 23182527
- [Background] Rudolph JL, Ramlawi B, Kuchel GA, McElhaney JE, Xie D, Sellke FW, Khabbaz K, Levkoff SE, Marcantonio ER. Chemokines are associated with delirium after cardiac surgery. J Gerontol A Biol Sci Med Sci. 2008 Feb;63(2):184-9. doi: 10.1093/gerona/63.2.184. PMID 18314455
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Kalisvaart KJ, de Jonghe JF, Bogaards MJ, Vreeswijk R, Egberts TC, Burger BJ, Eikelenboom P, van Gool WA. Haloperidol prophylaxis for elderly hip-surgery patients at risk for delirium: a randomized placebo-controlled study. J Am Geriatr Soc. 2005 Oct;53(10):1658-66. doi: 10.1111/j.1532-5415.2005.53503.x. PMID 16181163
- [Background] Mu DL, Zhang DZ, Wang DX, Wang G, Li CJ, Meng ZT, Li YW, Liu C, Li XY. Parecoxib Supplementation to Morphine Analgesia Decreases Incidence of Delirium in Elderly Patients After Hip or Knee Replacement Surgery: A Randomized Controlled Trial. Anesth Analg. 2017 Jun;124(6):1992-2000. doi: 10.1213/ANE.0000000000002095. PMID 28525512
- [Background] Peng K, Liu HY, Wu SR, Cheng H, Ji FH. Effects of Combining Dexmedetomidine and Opioids for Postoperative Intravenous Patient-controlled Analgesia: A Systematic Review and Meta-analysis. Clin J Pain. 2015 Dec;31(12):1097-104. doi: 10.1097/AJP.0000000000000219. PMID 25654534
- [Derived] Hong H, Zhang DZ, Li M, Wang G, Zhu SN, Zhang Y, Wang DX, Sessler DI. Impact of dexmedetomidine supplemented analgesia on delirium in patients recovering from orthopedic surgery: A randomized controlled trial. BMC Anesthesiol. 2021 Sep 13;21(1):223. doi: 10.1186/s12871-021-01441-3. PMID 34517840